CLINICAL TRIAL: NCT03588494
Title: Recombinant Human Endostatin (Endostar) Combined With Concurrent Chemoradiotherapy for Advanced Non-small Cell Lung Cancer: A Multicenter, Randomized, Controlled Trial
Brief Title: Endostar in Combination With Chemoradiotherapy in Patient With Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Afﬁliated Hospital of North Sichuan Medical College (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, DaiYuan Ma, Director of Cancer Center, Afﬁliated Hospital of North Sichuan Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSOG001
Record Dates: First submitted 2018-06-23; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Quality of Life
Keywords: Recombinant human endostatin; NSCLC; chemoradiotherapy
MeSH Terms: interventions — Chemoradiotherapy; endostar protein

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to a regimen of W1-CCRT(one treatment cycle of intravenous pump of recombinant human endostatin before chemoradiotherapy), or W2-CCRT(two treatment cycle of intravenous pump of recombinant human endostatin before chemoradiotherapy), or CCRT.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- concurrent chemoradiotherapy (CCRT) (Active Comparator): Chemotherapy: Cisplatin (50 mg/m2) on days 1, 8, 29, and 36 and etoposide (50mg/m2) on days 1～5 and 29～33.
  Radiotherapy: Thoracic radiotherapy (TRT) started with a linear accelerator (6MV-X) on the first day of chemotherapy.A minimum dose of 60 Gy (2 Gy per fraction, Monday～Friday) was delivered, and a range of 60-66 Gy in 2 Gy fractions was allowed.
  Interventions: Combination Product: concurrent chemoradiotherapy (CCRT)
- W1-CCRT (Experimental): Endostar(15 mg/m2) was durative transfused every 24 hours for 5 days during the normalization window of the first chemoradiotherapy cycle(days -5～-1).
  Chemotherapy: Cisplatin (50 mg/m2) on days 1, 8, 29, and 36 and etoposide (50mg/m2) on days 1～5 and 29～33.
  Radiotherapy: Thoracic radiotherapy (TRT) started with a linear accelerator (6MV-X) on the first day of chemotherapy.A minimum dose of 60 Gy (2 Gy per fraction, Monday～Friday) was delivered, and a range of 60-66 Gy in 2 Gy fractions was allowed.
  Interventions: Combination Product: concurrent chemoradiotherapy (CCRT); Drug: Endostar for one cycle
- W2-CCRT (Experimental): Endostar(15 mg/m2) was durative transfused every 24 hours for 5 days during the normalization window of the first and the second chemoradiotherapy cycles(days -5～-1 and 24～28).
  Chemotherapy: Cisplatin (50 mg/m2) on days 1, 8, 29, and 36 and etoposide (50mg/m2) on days 1～5 and 29～33.
  Radiotherapy: Thoracic radiotherapy (TRT) started with a linear accelerator (6MV-X) on the first day of chemotherapy.A minimum dose of 60 Gy (2 Gy per fraction, Monday～Friday) was delivered, and a range of 60-66 Gy in 2 Gy fractions was allowed.
  Interventions: Combination Product: concurrent chemoradiotherapy (CCRT); Drug: Endostar for two cycles

INTERVENTIONS:
Combination Product: concurrent chemoradiotherapy (CCRT) — Chemotherapy: Cisplatin (50 mg/m2) on days 1, 8, 29, and 36 and etoposide (50mg/m2) on days 1～5 and 29～33.
  Radiotherapy: Thoracic radiotherapy (TRT) started with a linear accelerator (6MV-X) on the first day of chemotherapy.A minimum dose of 60 Gy (2 Gy per fraction, Monday～Friday) was delivered, and a range of 60-66 Gy in 2 Gy fractions was allowed.
Drug: Endostar for one cycle — Endostar(15mg/m2) was durative transfused during the normalization window of the first chemoradiotherapy cycle(days -5～-1).
  Arms: W1-CCRT
Drug: Endostar for two cycles — Endostar(15mg/m2) was durative transfused during the normalization window of the first and the second chemoradiotherapy cycles(days -5～-1 and 24～28).
  Arms: W2-CCRT

SUMMARY:
To investigate the safety and efficacy recombinant human endostatin(endostar) durative transfusion combined with cocurrent chemoradiotherapy in advanced non-small cell lung cancer(NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients, age: 18-70 years of age
* 2. Pathology was diagnosed as non-small cell lung cancer. According to the Tumor Node Metastasis（TNM）stage of the 8th edition of the International Association for the Study of Lung Cancer in 2017, And the pathological stage was identified as stage IIIa-b.
* 3. No previous chest radiotherapy and radiotherapy, immunotherapy or biological therapy.
* 4. Eastern Cooperative Oncology Group (ECOG) test scored 0-1.
* 5. Serum hemoglobin ≥ 100g/L, platelet ≥ 100 × 109/L, absolute number of neutrophils ≥ 1.5 × 109/L.
* 6. Serum creatinine ≤ 1.25 times the upper limit of normal(UNL) or creatinine clearance ≥ 60 mL/min.
* 7. Serum bilirubin ≤ 1.5 times UNL, Aspartate aminotransferase (AST) and adenosine triphosphate (ALT) ≤ 2.5 times UNL, alkaline phosphatase ≤ 5 times UNL.
* 8. Forced vital capacity rate of one second（FEV1）>0.8 litre.
* 9. Coagulation function is normal
* 10. lesions are measurable according to the Response Evaluation Criteria in Solid Tumors Version 1.1(RECIST1.1)standard
* 11. Sign the inform consent form with good compliance

Exclusion Criteria:

* 1. Carcinoid or small cell lung cancer
* 2. Patients with any distant metastasis
* 3. patients with previous or current malignancy, except for skin non-melanoma or carcinoma in situ in the cervix
* 4. Any other disease or condition is a contraindication to chemoradiation (eg, active infection, 6 months after myocardial infarction, symptomatic heart disease including unstable angina, congestive heart failure or uncontrolled arrhythmia, immunosuppressive therapy).
* 5. Pregnancy or breastfeeding women
* 6. Women who may be pregnant but are unwilling to take appropriate contraception
* 7. Hereditary bleeding or coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 4 years
  Evaluate the effect of chemoradiotherapy with or without recombinant human endostatin on progression free survival

SECONDARY OUTCOMES:
Overall Survival(OS) | 4 years
  comparison to maintenance chemoradiotherapy alone
Treatment-related toxicity | 4 years
  Toxicity and adverse events related to the inventions

CONTACTS AND LOCATIONS:
Overall Officials: Daiyuan Ma, M.D, Principal Investigator — Afﬁliated Hospital of North Sichuan Medical College
Locations (1):
- Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided